CLINICAL TRIAL: NCT03485833
Title: End-expiratory and End-inspiratory Occlusion Tests to Predict Fluid Responsiveness in Mechanically Ventilated Cardiac Surgical Patients
Brief Title: End-expiratory and End-inspiratory Occlusion Tests to Predict Fluid Responsiveness
Acronym: EEOFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EEOFR
Record Dates: First submitted 2018-03-24; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Surgery
Keywords: end-expiratory occlusion test; end-inspiratory occlusion test; transesophageal echocardiography; passive legs raising; fluid challenge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEO and EIO test (Experimental): velocity time integral of the aorta measured by transesophageal echocardiography during end expiratory and end inspiratory occlusion test to predict volume responsiveness.Responders are defined by an increase in velocity time integral over 15% after infusion of 5ml/kg of crystalloid solution.
  Interventions: Diagnostic Test: EEO and EIO test

INTERVENTIONS:
Diagnostic Test: EEO and EIO test — velocity time integral of the aorta measured by transesophageal echocardiography after end-expiratory and end-inspiratory occlusion test

SUMMARY:
The purpose of the study is to verify the efficacy of using end-expiratory and end-inspiratory occlusion tests as an index of fluid responsiveness in mechanically ventilated patients with cardiac surgery.

DETAILED DESCRIPTION:
Patients with hypotension after anesthetic induction for cardiac surgery, who requires fluid resuscitation based on clinical judgement by the anesthesiologists are enrolled in this study. Patients are monitored by transesophageal echocardiography and FloTrac/Vigileo. Hemodynamic variables (heart rate, systolic blood pressure, diastolic blood pressure, mean artery pressure, central venous pressure, stroke volume variation, cardiac index, velocity time integral of the aorta etc) are measured at baseline, after end-expiratory occlusion (EEO) test, after end-inspiratory occlusion (EIO) test, after passive legs raising test, and after fluid challenge respectively. Responders are defined by an increase in velocity time integral over 15% after infusion of 5ml/kg of crystalloid solution.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgical patients
* hypotension after induction of anesthesia
* required volume expansion by clinical judgement of the anesthesiologist

Exclusion Criteria:

* younger than 18 years
* severe valve regurgitation or systolic dysfunction of the right ventricle
* contraindication of the transesophageal echocardiography examination
* cardiac arrhythmia
* left ventricular ejection fraction less than 30% before surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
responders | within 1 minute after volume expansion
  responders are defined by volume time integral increases over 15% after volume expansion of 5ml/kg crystalloid

SECONDARY OUTCOMES:
nonresponders | within 1 minute after volume expansion
  nonresponders are defined by volume time integral increases less than 15% after volume expansion of 5ml/kg crystalloid

CONTACTS AND LOCATIONS:
Overall Officials: Guo-wei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No